CLINICAL TRIAL: NCT02923609
Title: A PILOT TRIAL OF CELL THERAPY IN HEART FAILURE WITH PRESERVED EJECTION FRACTION
Brief Title: Cell Therapy in HFpEF
Acronym: CELLpEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Bojan Vrtovec, Medical Director, Advanced Heart Failure and Transplantation Programme, University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CELLpEF
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure With Normal Ejection Fraction
MeSH Terms: interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Intervention Model Description: The study is designed in a prospective crossover fashion. In Phase 1 of the study, all patients are treated with optimization of medical therapy for 6 months. Thereafter, all patients cross over to Phase 2 of the study, where they receive transendocardial CD34+ cell therapy. Follow-up of Phase 2 lasts for 6 months. At the time of enrollment (6 months before cell therapy), at time of cell therapy, and 6 months thereafter we will perform detailed clinical evaluation, laboratory assays, echocardiography, 6-minute walk test, and measure plasma levels of N-terminal pro B-type natriuretic peptide (NT-proBNP).
Masking Description: The echocardiographer will be blinded for the timing of echocardiographic recordings.
Oversight: Data Monitoring Committee: No

ARMS (1):
- SC Group (Experimental): In Phase 1 of the study, all patients will be treated with optimization of medical therapy for 6 months. Thereafter, all patients will cros over to Phase 2 of the study, where they will receive transendocardial CD34+ cell therapy. Follow-up of Phase 2 will last for 6 months. At the time of enrollment (6 months before cell therapy), at time of cell therapy, and 6 months thereafter we will perform detailed clinical evaluation, laboratory assays, echocardiography, 6-minute walk test, and measure plasma levels of N-terminal pro B-type natriuretic peptide (NT-proBNP).
  Interventions: Biological: Cell Therapy

INTERVENTIONS:
Biological: Cell Therapy — Electro-anatomical mapping will be performed using the Biosense NOGA system (Biosense-Webster, Diamond Bar, California). Local diastolic function will be assessed by a novel algorhithm that allows for the measuring local ventricular relaxation times at each of the sampling points. Target areas for cell delivery will be defined as the myocardial segments with the evidence of local diastolic dysfunction and myocardial hibernation. Transendocardial delivery of cell suspension in the SC Group will be performed with MyoStar® (Biosense Webster) injection catheter. Each patient will receive 20 injections of 0.3 mL of stem cell suspension.

SUMMARY:
The primary objective of the study is to investigate safety and efficacy of transendocardial CD34+ cell therapy in patients with HFpEF by evaluating changes in myocardial structure and function, patient exercise capacity and clinical outcome.

The safety end-points include serious adverse events (SAEs), defined as any serious event that may result in persistent or significant disability or incapacity and included death, heart transplantation, sustained ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation), and heart failure exacerbation requiring hospitalization.

DETAILED DESCRIPTION:
In all patients, peripheral blood stem cells will be mobilized by daily subcutaneous injections of G-CSF (10 mcg/kg, divided b.i.d) for 5 days. Peripheral blood stem cells will then be collected with Miltenyi cell separator (Miltenyi Biotech, Germany) and the magnetic cell separator Isolex 300i (Nexell Therapeutics Inc., California, USA) will be used for the immunomagnetic positive selection of the CD34+ cells.

ELIGIBILITY:
Inclusion Criteria:

* Preserved left ventricular systolic function on echocardiography (LVEF>50%)
* Evidence of diastolic dysfunction by echocardiography (E/e'>15)
* Symptoms of heart failure
* NT-proBNP levels >300 pg/ml
* absence of permanent atrial fibrillation

Exclusion Criteria:

* acute multi-organ failure
* history of any malignant disease within 5 years
* diminished functional capacity due to non-cardiac co-morbidities (COPD, PAOD, morbid obesity)
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular filling pressures (E/e') assessed by echocardiography | Baseline, 6 months and 1 year
  The E/e' ratio will be calculated from early transmitral velocity divided by peak left ventricular relaxation velocity for estimation of the left ventricular filling pressure.

SECONDARY OUTCOMES:
Change in exercise capacity | Baseline, 6 months and 1 year
  6-minute walk test will be performed by a blinded observer according to the standard protocol.
Change in NT-proBNP levels | Baseline, 6 months and 1 year
  NT-proBNP assays will be performed at a central independent laboratory, blinded to the patient's clinical data using a commercially available kit (Roche Diagnostics, Mannheim, Germany).
Change in systolic strain | Baseline, 6 months and 1 year
  Left ventricular longitudinal strains will be analyzed by speckle tracking echocardiography from apical four-chamber, two-chamber, and long-axis views.
Change in diastolic dysfunction grade | Baseline, 6 months and 1 year
  Diastolic dysfunction will be graded according based on E/A ratio and left atrial pressure estimation.

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Vrtovec, MD, PhD, Principal Investigator — Department of Cardiology, UMC Ljubljana
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vrtovec B, Frljak S, Poglajen G, Zemljic G, Cerar A, Sever M, Haddad F, Wu JC. A pilot clinical trial of cell therapy in heart failure with preserved ejection fraction. Eur J Heart Fail. 2022 Aug;24(8):1441-1449. doi: 10.1002/ejhf.2596. Epub 2022 Jul 20. PMID 35775390